CLINICAL TRIAL: NCT02458560
Title: Safety and Performance Study of the Edwards CENTERA-EU Self-Expanding Transcatheter Heart Valve
Brief Title: CENTERA-2: Safety and Performance Study of the Edwards CENTERA-EU Self-Expanding Transcatheter Heart Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Collaborators: Medstar Health Research Institute (Other); European Cardiovascular Research Center (Network); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-03
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Aortic Valve Disease
Keywords: Transcatheter Aortic Valve Replacement; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- single-arm (Experimental)
  Interventions: Device: Edwards CENTERA Self-Expanding Transcatheter Heart Valve

INTERVENTIONS:
Device: Edwards CENTERA Self-Expanding Transcatheter Heart Valve — The Edwards CENTERA Transcatheter Heart Valve (THV) System is indicated for use in symptomatic patients (high surgical risk) with severe aortic stenosis requiring aortic valve replacement (AVR).
  Other Names: TAVR; TAVI

SUMMARY:
The purpose of this study is to assess the safety and device success of the Edwards CENTERA Transcatheter Heart Valve (THV) System in symptomatic adult patients with severe aortic stenosis.

DETAILED DESCRIPTION:
This is a non-randomized, prospective, multi-center safety and device success study. Up to two hundred (200) patients are planned to be implanted at up to 35 participating investigational centers in Europe, Australia and New Zealand. Patient participation will last for a minimum of 5 years. Patients will be assessed at the following intervals: baseline, discharge, 30 days, 6 months, 1 year and annually thereafter through 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Heart team (including cardiac surgeon) agrees on eligibility including as-sessment that TAVI is appropriate.
2. High surgical risk: 8 ≤ STS Score ≤ 15 or 15 ≤ Logistic EuroSCORE I ≤ 40.
3. NYHA ≥ II.
4. Study patient is an adult of legal consent age.
5. Study patient has provided written informed consent to comply with all of the study procedures and follow-up visits.

Exclusion Criteria:

1. Acute myocardial infarction ≤ 30 days before the intended treatment.
2. Untreated clinically significant coronary artery disease requiring revascularization.
3. Aortic valve is a congenital unicuspid or congenital bicuspid valve.
4. Mixed aortic valve disease (with predominant aortic regurgitation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rate | 30 days post-index procedure

SECONDARY OUTCOMES:
Safety composite of mortality, stroke, major vascular, complication, life-threatening bleeding, acute kidney injury coronary artery obstruction requiring intervention, and THV-related dysfunction requiring repeat procedure. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Windecker, MD, Principal Investigator — Inselspital Bern (Switzerland); Prof. Hermann Reichenspurner, MD, Principal Investigator — University Heart Center Hamburg (Germany)
Locations (27):
- Australia (3):
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Epworth Healthcare, Melbourne, Victoria
- Rigshospitalet, Copenhagen, Denmark
- France (3):
  - Institut Hospitalier Jacques Cartier, Massy
  - CHU Pontchaillou, Rennes
  - Clinique Pasteur, Toulouse
- Germany (11):
  - Klinikum Augsburg, Augsburg
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Charité - Universitaetsmedizin Berlin, Berlin
  - Herzzentrum Universitaet Bonn, Bonn
  - Asklepios Klinik St Georg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Staedtisches Klinikum Karlsruhe GmbH & Helios Herzchirurgie Karlsruhe GmbH, Karlsruhe
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum Muenchen, Munich
  - LMU - Klinikum der Universitaet Muenchen, Munich
  - Universitaetsklinikum Muenster, Münster
- Italy (3):
  - Ospedale Ferrarotto - Azienda Ospedaliero Universitaria di Catania, Catania
  - Ospedale San Raffaele s.r.l., Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
- Netherlands (3):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - Universitair Medical Center (UMC) Utrecht, Utrecht
- Auckland City Hospital, Grafton, Auckland, New Zealand
- Inselspital Bern, Bern, Switzerland
- Royal Victoria Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tchetche D, Windecker S, Kasel AM, Schaefer U, Worthley S, Linke A, Abdel-Wahab M, Le Breton H, Sondergaard L, Spence MS, Petronio S, Baumgartner H, Hovorka T, Blanke P, Reichenspurner H. 1-Year Outcomes of the CENTERA-EU Trial Assessing a Novel Self-Expanding Transcatheter Heart Valve. JACC Cardiovasc Interv. 2019 Apr 8;12(7):673-680. doi: 10.1016/j.jcin.2019.01.231. PMID 30947942
- [Derived] Reichenspurner H, Schaefer A, Schafer U, Tchetche D, Linke A, Spence MS, Sondergaard L, LeBreton H, Schymik G, Abdel-Wahab M, Leipsic J, Walters DL, Worthley S, Kasel M, Windecker S. Self-Expanding Transcatheter Aortic Valve System for Symptomatic High-Risk Patients With Severe Aortic Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3127-3136. doi: 10.1016/j.jacc.2017.10.060. PMID 29268926